CLINICAL TRIAL: NCT06075316
Title: Improving Thoracic Surgical Care Using Electronic Patient-Reported Outcomes (ePROS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LCCC 2141; 1K23HL157765-01A1 (NIH)
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Thoracic
Keywords: Electronic Patient-Reported Outcome; Patient-Reported Outcome; thoracic surgery; complications

STUDY DESIGN:
Intervention Model Description: The participants will have their alerts sent to the clinicians when concerning symptoms are reported.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ePRO monitoring (Other): Thoracic surgery patients will be enrolled in ePRO monitoring using web-based or telephone surveys.
  Interventions: Other: Symptom monitoring

INTERVENTIONS:
Other: Symptom monitoring — Alerts will be sent to providers via email and/or the electronic medical record at pre-specified response thresholds. Providers will be instructed to respond to and document the management of alerts per their clinical routine.

SUMMARY:
This is a single-site, non-randomized study on the outcomes of remote real-time "ePRO monitoring" in thoracic surgery patients. ePRO monitoring is a health information technology intervention comprised of delivering longitudinal electronic patient-reported outcome (ePRO) surveys (e.g., on symptoms, and physical functioning) coupled with automated provider alerts for concerning survey responses.

DETAILED DESCRIPTION:
Thoracic surgery patients are at high risk for severe complications post-surgery, such as respiratory failure, empyema, wound problems, and even mortality. Patients with complications may need readmission and invasive management. Usual care may not capture the symptoms of surgery complications. Well-designed remote monitoring of postoperative patients may enable early intervention and lower the risk of severe complications.

This study evaluates the implementation and effectiveness of perioperative electronic patient-reported outcomes (ePROs) monitoring in thoracic surgery patients. Previous studies demonstrated the feasibility of ePROs monitoring by thoracic surgery patients and providers. This study will explore barriers to implementation before real-world effectiveness studies.

ELIGIBILITY:
Inclusion Criteria:

Patients participating in ePRO monitoring must meet the following inclusion criteria to participate in this study:

1. 18 years or older
2. English or Spanish speaking
3. Able to complete a web-based, telephonic (IVR), or CRA (or other IRB-approved research team member)-administrated symptom survey
4. Planned to undergo major thoracic surgery (involving chest wall incisions and overnight admission)
5. Discharged from the thoracic surgery service
6. Discharged to home

Exclusion Criteria:

All patients meeting any of the following exclusion criteria at enrollment will be excluded from study participation:

1. Not completing planned surgery within 3 months of obtaining informed consent
2. Inability to understand English or Spanish
3. Having undergone only minor thoracic surgery (e.g. bronchoscopy, cervical mediastinoscopy)
4. Dementia, altered mental status, or any psychiatric condition determined by the thoracic surgery provider team that would prohibit the understanding or rendering of informed consent.
5. Current incarceration
6. Pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Reach of ePRO monitoring | Months 4 through 6 after implementation of the study
  Percentage of eligible thoracic surgery patients enrolling in ePRO monitoring.
Adoption of ePRO monitoring | Months 4 through 6 after implementation of the study
  Percentage of ePRO monitoring alerts sent that result in clinical action by providers within 1 week of delivery
Patient-level Uptake | Months 4 through 6 after implementation of the study
  the percentage of enrolled patients who participate in >=1 ePRO survey.
Overall Reach of ePRO monitoring | End of study
  Percentage of eligible thoracic surgery patients enrolling in ePRO monitoring.

SECONDARY OUTCOMES:
Complication Rate | Baseline through 30 days post-discharge
  Percentage of participants with severe complications (Clavien-Dindo grade >=3)
Emergency department visit at 30 days | Baseline through 30 days post-discharge
  Percentage of participants with an emergency department visit
Emergency department visit at 90 days | Baseline through 90 days post-discharge
  Percentage of participants with an emergency department visit
Readmission at 30 days | Baseline through 30 days post-discharge
  Percentage participants readmitted to a hospital
Readmission at 90 days | Baseline through 90 days post-discharge
  Percentage participants readmitted to a hospital
Mortality at 30 days | Baseline through 30 days
  Percentage participants who died
Mortality at 90 days | Baseline through 90 days
  Percentage participants who died
Patient Alert Rate | Baseline through 90 days
  Percentage of all patients who trigger at least 1 alert.
Alert Rate | Baseline through 90 days
  Percentage of all ePRO surveys that trigger an alert

CONTACTS AND LOCATIONS:
Overall Officials: Gita Mody, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plan as of now to make IPD available to other researchers.

REFERENCES:
- See also: Clinical trials at UNC Lineberger — http://unclineberger.org/patientcare/clinical-trials/clinical-trials